CLINICAL TRIAL: NCT00694031
Title: A Randomized Study to Evaluate Survival in Patients Undergoing Hemodialysis or On-line Hemodiafiltration
Brief Title: Survival Study in Patients Undergoing On-line Hemodiafiltration
Acronym: ESHOL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Societat Catalana de Nefrologia (Unknown)
Responsible Party: Principal Investigator, Francisco Maduell, Dr, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESHOL
Record Dates: First submitted 2008-06-05; First posted 2008-06-10 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2012-06

CONDITIONS: Hemodialysis
Keywords: Mortality; Convective therapies; On-line Hemodiafiltration; Dialysis Adequacy; Age 18 or older; Undergoing hemodialysis
MeSH Terms: interventions — Renal Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Hemodialysis
  Interventions: Procedure: Hemodialysis
- B (Experimental): On-line hemodiafiltration
  Interventions: Procedure: On-line hemodiafiltration

INTERVENTIONS:
Procedure: Hemodialysis — 3 times per week
  Arms: A
Procedure: On-line hemodiafiltration — 3 times per week
  Arms: B

SUMMARY:
Patients on hemodialysis will be randomly assigned (1:1) to continue on conventional hemodialysis or on-line hemodiafiltration, both three times per week. A 3 year follow-up and a sample size of around 750 will be necessary to detect a 35% reduction in mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Currently undergoing hemodialysis
* Clinical stability
* Stable vascular access

Exclusion Criteria:

* Chronic inflammatory diseases
* Liver cirrhosis
* Malignancies
* Chronic immunosuppressant or antiinflammatory use
* Dialysis through temporary catheter or single puncture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 906 (Actual)
Dates: Start 2007-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Survival | 36 months

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Clinic de Barcelona, Barcelona, Barcelona
  - CSU Bellvitge, L'Hospitalet de Llobregat, Barcelona

REFERENCES:
- [Background] Maduell F, Moreso F, Pons M, Ramos R, Mora-Macia J, Foraster A, Soler J, Galceran JM, Martinez-Castelao A; Online Hemodiafiltration Study Group from the Catalonian Society of Nephrology. Design and patient characteristics of ESHOL study, a Catalonian prospective randomized study. J Nephrol. 2011 Mar-Apr;24(2):196-202. doi: 10.5301/jn.2010.386. PMID 20602331
- [Background] Maduell F, Moreso F, Pons M, Ramos R, Mora-Macia J, Carreras J, Soler J, Torres F, Campistol JM, Martinez-Castelao A; ESHOL Study Group. High-efficiency postdilution online hemodiafiltration reduces all-cause mortality in hemodialysis patients. J Am Soc Nephrol. 2013 Feb;24(3):487-97. doi: 10.1681/ASN.2012080875. Epub 2013 Feb 14. PMID 23411788